CLINICAL TRIAL: NCT05994924
Title: A Pilot Randomized Controlled Trial Using Storytelling To Prevent Obesity and Encourage Responsive Feeding Practices in Young Children
Brief Title: Storytelling To Prevent Obesity and Encourage Responsive Feeding Practices in Young Children
Acronym: STORY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00078071
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-05

CONDITIONS: Obesity, Childhood
Keywords: obesity; young children; feeding practices; obesity prevention; obesity intervention; child feeding questionnaire; satiety responsiveness; food responsiveness; family meal frequency questionnaire; structure of family meals
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Handout Only (Active Comparator): Parents in this group receive an educational handout at the baseline visit.
  Interventions: Behavioral: Educational Handout
- Online-Only Video Series (Active Comparator): Parents will be given (QR) quick-response codes to watch the videos on their own time with no discussion afterward.
  Interventions: Behavioral: Video Series
- Group Sessions (Active Comparator): Parents will participate in 2 weekly group sessions with video viewing and group discussion.
  Interventions: Behavioral: Video Series; Behavioral: Group Discussion Sessions

INTERVENTIONS:
Behavioral: Educational Handout — Educational handout describing responsive feeding practices.
  Arms: Handout Only
Behavioral: Video Series — Videos geared toward responsive feeding practices.
  Arms: Group Sessions; Online-Only Video Series
Behavioral: Group Discussion Sessions — Group discussion following video viewing led by Imprints Cares, a community organization focused on early childhood education.
  Arms: Group Sessions

SUMMARY:
The goal of this qualitative trial study is to assess the usefulness and acceptability of the intervention in diverse clinical and community settings. The main questions it aims to answer are:

* How many parents were approached and consented to participate?
* How many parents viewed the videos via link versus viewed the video with a discussion in group sessions?
* How did parents feel about the process of being recruited and interventions that they participated in?
* How did the providers feel about the intervention recruitment and delivery?
* How did the facilitators feel about their delivery of the material? Participants will complete a survey and an interview after completing second part of the intervention.

Researchers will compare handout, online-only video, and group class interventions to see if an intervention delivery is useful and accepted by parents or providers.

DETAILED DESCRIPTION:
This is a pilot randomized trial to assess feasibility and acceptability of STORY. The study will recruit 30 parents. Parents will complete a questionnaire and dyad's heights and weights will be measured. Families will be randomized to the control group or 1 of 2 intervention delivery approaches (IA). Parents will be given a handout (controls), links to the videos to watch independently (IA 1), or information on how they will be contacted to schedule their intervention sessions (IAs 2). After 2 video/sessions, all parents will complete a written survey assessing their experience with the intervention and any change same at home; the written survey will reassess baseline measures. Intervention parents will also complete a semi-structured interview to assess the family's experience with the STORY trial.

Sub aim 2a: Feasibility: number of parents approached, number of parents consented Sub aim 2b: Adherence: number of parents who complete videos or sessions Sub aim 2c: Acceptability to parents and providers

ELIGIBILITY:
Inclusion Criteria:

* Parent of 2-4 year old child
* Is at least 18 years old
* Participant can read and write English
* The participant's child has no medical conditions that affect development, feeding, or growth

Exclusion Criteria:

* Participant is not a parent of a 2-4 year old child
* Parent is less than 18 years old
* Parent can not read and write English
* Participant's child has a medical condition that affects development, feeding, or growth
* Family/household member participating in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Number of Parents Approached | Baseline
  Number of parents who are approached for participation at 3 primary care offices.
Number of Parents Consented | Baseline
  Number of parents that consented to participating in the study.
Number of Parents who Viewed Videos Provided by Provider | Month 2
  tracking the number of videos viewed by each parent
Number of Parents who Complete In-Person Group Sessions | Month 2
  tracking the number of sessions attended by each parent
Parent Acceptance of Intervention - Percent of parents | Month 4
  Measure parent acceptability of intervention using brief survey and semi-structured interview responses - Percent of parents who respond on the survey that the intervention was acceptable or completely acceptable to them
Provider Acceptance of Intervention - Percent of providers | Month 4
  Measure provider acceptability using a short survey - Percent of providers who respond on the survey that the intervention was acceptable or completely acceptable to them
Facilitator Acceptance of Intervention - Percent of facilitators | Month 4
  Measure facilitator acceptability using semi-structured interviews - Percent of facilitators who respond on the survey that the intervention was acceptable or completely acceptable to them

SECONDARY OUTCOMES:
Mean pressure to eat score (Child Feeding Questionnaire) | Month 4
  The 4-item subscale from the Child Feeding Questionnaire, called Pressure to Eat, measures parents' tendency to pressure their children to eat more food, typically at mealtimes. Possible scores range from 1-5, with higher scores indicating greater severity of parents' tendency to pressuring their children to eat more food. Information to be utilized in a future larger study.
Mean restriction score (Child Feeding Questionnaire) | Month 4
  The 8-item subscale from the Child Feeding Questionnaire, called Restriction, measures the extent to which parents restrict their child's access to foods. Possible scores range from 1-5, with higher scores indicating greater severity of parents restricting their child's access to foods. Information to be utilized in a future larger study.
Mean satiety responsiveness score | Month 4
  Mean satiety responsiveness score obtained using a 5-point scale from Child Eating Behavior Questionnaire. Possible scores range from 1-5, with higher scores indicating higher self-regulation. Information to be utilized in a future larger study.
Mean food responsiveness score | Month 4
  Mean food responsiveness score obtained using a 5-point scale from Child Eating Behavior Questionnaire. Possible scores range from 1-5, with higher scores on food responsiveness indicating lower self-regulation. Information to be utilized in a future larger study.
Mean enjoyment of food score | Month 4
  Mean enjoyment of food score obtained using a 5-point scale from Child Eating Behavior Questionnaire. Possible scores range from 1-5, with higher scores on food responsiveness indicating lower self-regulation. Information to be utilized in a future larger study.
Mean of families using structured mealtime practices | Month 4
  The 10-item Structure of Family Meals subscale from the Meals in our Household Questionnaire measures how often families spend their mealtimes in a specific setting. Possible scores range from 0-4, with higher scores indicating higher occurrences of specific mealtime settings. Information to be utilized in a future larger study.
Percentage of families eating family meals at least 3 times per week | Month 4
  Percentage of families eating family meals at least 3 times per week using Family Meal Frequency Questionnaire which asks how many times a week the family eats dinner together, both at home and at a restaurant. Information to be utilized in a future larger study.
Percentage of Parents that are categorized into four feeding styles (Caregiver's Feeding Styles Questionnaire Reduced Version) | month 4
  The 10-item questionnaire is measured on a 5-point Likert scale (ranging from 1=never to 5=always). The demandingness and responsiveness scores are used to categorize parent feeding style into one of four categories: authoritative, authoritarian, indulgent, and uninvolved styles.
Fidelity of intervention delivery - Percentage of key points | month 4
  Study staff will complete Evaluation Checklist of key points communicated during each session to determine intervention delivery - Percentage of key points communicated during the sessions from the Evaluation Checklist
Facilitator Self-Competence Percentage - Percentage of facilitators | month 4
  Facilitator self-competence percentage will be collected from facilitators responding to an open-ended question after each session to evaluate the strong and weak points of their own delivery - : Percentage of facilitators who respond agree or strongly agree to survey question about perceived self-competence
Fidelity of Receipt - : Percentage of parents | month 4
  Percentage of parents who respond agree or strongly agree to survey question about whether the video content was relevant
Percentage of Parents who Identified a Goal | month 4
  Receipt will be collected through the follow-up survey. Information collected includes a response of "yes" or "no" by parent expert assessment of whether the parent identified an attainable, specific, and measurable goal. Percentage of parents who identified a goal will include the percentage who answer "yes".
Enactment percentage | month 4
  Enactment will be collected through the follow-up survey. Enactment Percentage will include those considered by an expert to have made a specific and measurable change in feeding practices.

OTHER OUTCOMES:
Qualitative Analysis | month 4
  Information collected from semi-structured interviews. Thematic analysis performed and coded by two independent investigators. Representative quotes will be recorded, and transcript codes will be grouped into similar categories. Investigators will interpret themes and sub-themes from these categories.

CONTACTS AND LOCATIONS:
Overall Officials: Callie Brown, MD, MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT05994924/Prot_SAP_001.pdf
  • Informed Consent Form (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT05994924/ICF_000.pdf